CLINICAL TRIAL: NCT05053165
Title: A Phase 1, Randomised, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of LB-P6 or LB-P8 in Healthy Participants
Brief Title: A Study to Assess the Safety and Tolerability of LB-P6 and LB-P8 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LISCure Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB-001
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis; Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (LB-P6) (Experimental): Healthy volunteers will be administered once daily orally
  Interventions: Drug: LB-P6
- B (LB-P8) (Experimental): Healthy volunteers will be administered once daily orally
  Interventions: Drug: LB-P8
- C (Placebo) (Experimental): Healthy volunteers will be administered once daily orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB-P6 — Healthy subjects will be randomized to receive LB-P6 once daily orally
  Arms: A (LB-P6)
Drug: LB-P8 — Healthy subjects will be randomized to receive LB-P8 once daily orally
  Arms: B (LB-P8)
Drug: Placebo — Healthy subjects will be randomized to receive placebo once daily orally
  Arms: C (Placebo)

SUMMARY:
The study is designed to assess the safety and tolerability of multiple ascending doses of LB-P6 or LB-P8 in healthy participants.

DETAILED DESCRIPTION:
This is randomised, double-blind, placebo-controlled, single centre study to assess the safety and tolerability of multiple ascending doses of LB-P6 or LB-P8 in healthy participants.

A total of up to 30 healthy participants will be enrolled in 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 65 years (inclusive at the time of consent).
2. BMI ≥ 18 to ≤ 32 kg/m2 and with weight ≥ 50 kg at Screening.
3. Must have a negative urine drug screen at the Screening Visit and the day before dosing (Day -1); one repeat urine drug may be conducted for a suspected false positive result.
4. Female participants should meet 1 of the following criteria before they can participate in the study:

   1. Not of childbearing potential, defined as surgically sterile for at least 12 months prior to screening or postmenopausal
   2. Of childbearing potential and agrees to take effective contraceptive measures throughout the study period from study entry (ie, screening) until at least 3 months after the last dose of IP.
   3. Of childbearing potential and in an exclusive relationship with a partner who has had a bilateral vasectomy at least 6 months prior to study entry.

   Female participant of childbearing potential must have a negative serum pregnancy test at Screening, and a negative urine pregnancy test at Baseline (ie, Day -1), and be willing to have additional pregnancy tests, as required, throughout the study, at the discretion of the PI or designee.
5. Male participant: has undergone bilateral vasectomy (at least 6 months prior to study entry) or agrees to use effective contraceptive measures and not donate sperm throughout the study period from study entry (ie, Screening) until at least 3 months after the last dose of IP.
6. Must agree to adhere to the current state and national advice regarding minimising exposure to COVID-19 from the first Screening Visit until the EOS Visit.

Exclusion Criteria:

1. Female participants who are pregnant, lactating, or who plan to become pregnant within 90 days of the EOS Visit.
2. The participant has either a history or presence of any clinically significant immunological disorder/disease (such as autoimmune diseases, etc.), cardiovascular, thromboembolic events, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (particularly diabetes or prediabetes), haematological, dermatological, venereal, neurological, chronic infectious or psychiatric disease or other major disorder that, in the opinion of the PI or designee, may interfere with trial compliance, completion, or accurate assessment of trial outcomes or safety.
3. The participant has taken prescription (including antibiotics and anti-virals) or non prescription medication, herbal remedies, vitamins or minerals, any probiotics and yeast supplements within 14 days prior to the first dose of IP unless in the opinion of the PI or designee the medication will not compromise participant safety or interfere with study procedures or data validity. Participants may be rescreened after a washout period of 14 days. Use of contraceptives and paracetamol up to 2 g/day and/or nonsteroidal anti inflammatory drugs (NSAIDs) for symptomatic relief of minor symptoms are allowed.
4. The participant has a substance abuse-related disorder or has a history of drug, alcohol, and/or substance abuse deemed significant by the PI or designee. Any participant with a positive screen for drugs of abuse or alcohol at Screening or on Day -1 will also be excluded.
5. The participant has taken any IPs within 30 days prior to the first dose of IP or 5 half-lives, whichever is longer.
6. Positive test result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus antibody (anti-HCV), FOB at Screening.
7. The participant has a fever (body temperature > 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to admission to the clinical research unit (CRU).
8. The participant has undergone vaccination (including with a live-attenuated vaccine) within 30 days prior to Baseline (Day -1) through to the end of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending doses of LB-P6 or LB-P8 in healthy participants through adverse events as assessed by NCI-CTCAE v5.0 | Measurements at Baseline till 14 days after the last dose of study drug
  Number of participants with treatment related adverse events as assessed by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Cmax Clinical Research, Adelaide, Australia